CLINICAL TRIAL: NCT06851715
Title: Can the Quality of Life of Adolescents With Asthma be Improved by Focusing on Improving Their Asthma Self-management
Brief Title: Improving Quality of Life for Teenagers With Asthma
Acronym: IMPAQT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RHM CHI1258; 349662 (Other: Integrated Research Approval System (IRAS))
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Asthma in Children; Asthma
Keywords: Asthma; Adolescent; Self-efficacy; Quality of life; Asthma control
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinic consultation focused on asthma self-management (Experimental): The participant will complete the Adolescent Asthma Self-efficacy Questionnaire (AASEQ), and the clinic healthcare professional will use the responses to focus the consultation on areas where the participant needs support for asthma self-management.
  Interventions: Other: Clinic consultation focused on asthma self-management
- Usual clinic consultation (No Intervention): The participant will not complete the AASEQ at baseline and their healthcare professional will conduct the consultation as per usual management.

INTERVENTIONS:
Other: Clinic consultation focused on asthma self-management — The clinic healthcare professionals (HCPs) will be provided with the completed Adolescent Asthma Self-efficacy Questionnaire (AASEQ), which will help identify areas where participants need additional support to improve their asthma self-management skills. Targeted behavioural interventions, developed during the 'ItsMyAsthma' study, will be applied during the clinic consultation to address individual needs.
  Arms: Clinic consultation focused on asthma self-management

SUMMARY:
BACKGROUND: Asthma is a long-term lung condition affecting 1 in 11 children and young people in the UK. Many teenagers have well controlled asthma, but a significant number continue to experience regular symptoms and asthma attacks leading to hospitalisations. While non-adherence to medication is a factor, teenagers also face challenges like changing relationships with parents and peers, avoiding triggers like smoking, and fitting in treatment with daily life demands. Healthcare professionals (HCPs) also face difficulties in managing teenagers with asthma.

A previous study, funded by Asthma + Lung UK, developed a new approach to manage teenage asthma by focusing on self-efficacy, which is how confident one feels about performing a task. Teenagers completed the Adolescent Asthma Self-Efficacy Questionnaire (AASEQ), which identified areas where they needed more support. HCPs then tailored their consultations to address these needs. This approach improved the teenagers' confidence in self-managing their asthma.

Improving quality of life (QoL) is a key goal in asthma care. Therefore, the aim of this study is to determine if the self-efficacy approach improves QoL for teenagers with asthma.

METHODS: Teenagers aged 12-18 years with asthma will be recruited from hospital clinics. They will be randomly assigned to one of two groups:

1. Teenager will complete the AASEQ at the start of their appointment. The HCPs will use this to focus the consultation on areas where the teenager needs support in self-managing their asthma.
2. Teenager will have their usual consultation with the HCP.

Three months after the appointment, the QoL will be compared between the two groups using a standardised questionnaire.

IMPACT: If the self-efficacy approach proves to be beneficial, it could help HCPs to empower teenagers to better manage their asthma and ultimately improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent aged 12-18 years
* Attending a paediatric respiratory clinic
* Informed consent from adolescent aged ≥16 years, and assent plus parent/guardian consent for adolescents aged ≤16 years
* Paediatric Asthma Quality of Life Questionnaire score ≤5.5 points

Exclusion Criteria:

* Aged 0-11 or over 18 years
* Other significant long-term medical condition that has a day-to-day impact on their lives (except for co-existing allergic conditions, breathing pattern disorder, dysfunctional breathing, or intermittent laryngeal obstruction)
* Adolescent or parent/guardian unable to communicate sufficiently to complete consent forms.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Paediatric Asthma Quality of Life Questionnaire (PAQLQ) | 3 months after enrolment
  Paediatric Asthma Quality of Life Questionnaire score ranging from 0-36 points, with a higher score indicating worse quality of life.

SECONDARY OUTCOMES:
Asthma-related healthcare utilisation | 3 months after enrolment
  Asthma-related healthcare utilisation including number of asthma exacerbations requiring prednisolone/dexamethasone, and/or GP visits, Emergency Department, Hospital, or Intensive care admissions.
Asthma Control Test (ACT) | 3 months after enrolment
  Asthma Control Test score ranging from 5-25 points, with a higher score indicating better asthma control.
Adolescent Asthma Self-Efficacy Questionnaire (AASEQ) | 3 months after enrolment
  Adolescent Asthma Self Efficacy Questionnaire score ranging from 0-100 points, with a higher score indicating greater self-efficacy for management of asthma.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Rattu, Study Director — University of Southampton
Locations (2):
- United Kingdom (2):
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Isle of Wight NHS Trust, St Mary's Hospital, Isle of Wight, Isle of Wight

IPD SHARING:
Plan to Share IPD: Yes
Please contact the study investigators to request trial data. Note that it will need to be anonymised before sharing.